CLINICAL TRIAL: NCT06425614
Title: Centrifugation-based Versus Filtration-based Intraoperative Cell Salvage on Quality of Perioperative Haemostasis in Cardiac Surgery: A Randomized Clinical Trial
Brief Title: COmbined pLaTelet and eRythrocyte AutotransfusioN During Cardiac surgEry (COLTRANE) Trial
Acronym: COLTRANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHUBX 2022/22
Record Dates: First submitted 2024-01-12; First posted 2024-05-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: On-pump Cardiac Surgery; High Risk for Bleeding; Autotransfusion
Keywords: cardiac surgery; bleeding; autotransfusion; cardiopulmonary bypass; perioperative haemostasis; Universal Definition of Perioperative Bleeding; filtration-based autotransfusion; centrifugation-based autotransfusion
MeSH Terms: conditions — Hemorrhage | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Intervention Model Description: Multicentre clinical trial, Randomized, Comparative, controlled, single blinded, superiority design, two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autotransfusion by filtration (Experimental): new filtration-based autotransfusion (SAME I-SEP device)
  Interventions: Procedure: Autotransfusion
- Autotransfusion by centrifugation (Other): centrifugation-based autotransfusion (routinely used in cardiac surgery centers)
  Interventions: Procedure: Autotransfusion

INTERVENTIONS:
Procedure: Autotransfusion — ANTIFIBRINOLYTIC THERAPY :
  tranexamic acid as antifibrinolytic therapy : dose after anaesthesia induction followed by continuous intravenous infusion until end
  INTRAOPERATIVE MANAGEMENT :
  * Routine monitoring : five lead-ECG, pulse oximeter, non-invasive arterial pressure will be instituted. A peripheral venous catheter and an arterial catheter
  * The general anaesthesia :
  * propofol and Remifentanil or sufentanil both simultaneously administered .
  * monitoring of the bispectral index
  * Triple lumen central venous catheter
  * Heparinization (300 UI/kg)
  * Aortic and right auricular cannulations
  TRANSFUSION PROTOCOL :
  * During CPB, PRBC transfusion if necessary
  * In the postoperative period if necessary
  In bleeding patients:
  The perioperative use of blood products will be managed according to results of conventional haemostasis tests or viscoelastic point of care tests when available in the center.

SUMMARY:
Despite significant advances in patient blood management, cardiac surgery remains a surgical procedure at high risk for bleeding. Numerous perioperative blood conservation strategies have been developed for limiting the use of blood products. Among them, the processing of shed blood and residual cardiopulmonary bypass circuit volume with autotransfusion device is routinely used. Conventional centrifugation-based autotransfusion devices actually available only recover red blood cells while platelets and coagulation factors are almost totally lost. Consequently, large amounts of intraoperative cell salvage could significantly alter perioperative haemostasis. The SAME autotransfusion device (i-SEP, France) is a new and innovative filtration-based autotransfusion device able to recover erythrocytes, leukocytes but also platelets. By offering the opportunity to re-infuse to patients their own platelets in addition red blood cells, significantly improve perioperative haemostasis with this new device is expected. The purpose of the COLTRANE trial is to compare the quality of the perioperative haemostasis in cardiac surgical patients for whom intraoperative cell salvage will be performed using either the SAME autotransfusion device or conventional centrifugation-based device.

Because allogenic transfusion of blood products as well as surgical re-exploration for excessive bleeding are associated with poor outcomes and prolonged length of stay, the use of filtration-based SAME device by maintaining perioperative haemostasis could improve outcomes and reduce length of stay of high risk patients. The fact that patients receive their own platelets should also limit the risk of allo-immunization and immunomodulation which is recognized as one of the underlying mechanisms of perioperative increased risk of infection.

DETAILED DESCRIPTION:
The SAME device is a new and innovative filtration-based autotransfusion device able to recover both erythrocytes and platelets. A multicentre single-arm clinical feasibility and safety trial conducted by our group, using SAME device on 50 cardiac surgical patients reported erythrocyte yield per cycle of 89%, post-treatment hematocrit of 43% with an excellent washing performance. In addition, the device recovered 52% of platelets, that were found unaltered by the device as demonstrated by a limited platelet activation and a strong response to thrombin-pathway stimulation assessed by flow cytometry. By offering the opportunity to re-infuse to the patients their own platelets in addition to their RBC, this new device might significantly improve perioperative haemostasis and thus decrease the need for blood products. It is well established that severe postoperative bleeding and blood products transfusion lead to increase morbidity and mortality. Consequently, an improvement of postoperative outcomes and a decrease in intensive care unit (ICU) and hospital length of stay may be expected. The fact that patients receive their own platelets should limit the risk of allo-immunization and immunomodulation which is recognized as one of the underlying mechanisms of perioperative increased risk of infection. Consequently, a reduction of infectious complication may be also expected.

The purpose of COLTRANE trial is to test the hypothesis that the intraoperative use of the filtration-based SAME autotransfusion device could improve perioperative haemostasis thereby reducing the proportion of patients exhibiting clinically significant perioperative bleeding (moderate to massive bleeding according the Universal Definition of Perioperative Bleeding (UDPB) classification).

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 yr) affiliated or beneficiary of a social security scheme and undergoing on-pump cardiac surgery at high risk for bleeding with autotranfusion indication defined as:

* Primary or redo combined cardiac procedures (2 valves or more, valve(s) and coronary artery bypass grafting(s))
* Primary or redo ascending aorta surgery
* Primary or redo isolated coronary artery bypass grafting (iCABG) involving 3 or more grafts using the internal mammary artery
* Free, informed and written consent signed by the participant and the investigator

Exclusion Criteria:

* Preoperative therapy by P2Y12 receptor inhibitors (within 5 preoperative days for clopidogrel, ticagrelor or ticlopidine, within 7 preoperative days for prasugrel, and within one preoperative hour for cangrelor)
* Preoperative treatment by active anticoagulant drug (within 5 preoperative days for VKA, 4 days for dabigatran, 3 days for rivaroxaban and apixaban, 24 hours for therapeutic LMWH, 36 hours for therapeutic fondaparinux, 12 hours for prophylactic LMWH, 24 hours for prophylactic fondaparinux, 4 hours for unfractionated heparin Sepsis
* Malignant tumor
* Immunocompromised patients (steroids, immunosuppressive drugs, ongoing treatment for solid tumor or hematologic malignancy, primary immunodeficiency disorders, AIDS)
* Emergency cardiac surgery
* Heart transplantation
* Implantation or patients under ventricular assist device (VAD)
* Patients with two or more previous sternotomy
* Surgery procedure requiring circulatory arrest and/or profound hypothermia (<32°C)
* Active infective endocarditis
* Cardiac surgical procedure for benign or malignant cardiac tumors
* Patients with known acquired or constitutional coagulopathy requiring specialist management
* End stage renal disease
* Preoperative haemoglobin level less than 10 g/dL
* Preoperative platelet count < 100 G/L
* Persons participating in another interventional research including a period of exclusion that is still ongoing
* Pregnant or breastfeeding women
* Persons placed under judicial protection
* Patients deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Perioperative bleeding | At the end of Day 1
  The proportion of patients with clinically significant (moderate to massive) perioperative bleeding according to the Universal Definition for Perioperative Bleeding.

SECONDARY OUTCOMES:
total blood loss | Hours 12, Hours 24, up to 5 after operatives days
  Total blood loss from chest tubes within 12 and 24 postoperative hours and up to chest tubes removal (maximum 5 postoperative days)
surgical re-exploration | Day 0-Day 5,
  Surgical re-exploration for excessive bleeding within 5 postoperative days
Sternal closure | Hours 12
  Delayed sternal closure
Overall quality of perioperative haemostasis : Use of blood | Day 0-Day 2,
  Perioperative use of blood products and/or plasma derivatives within 2 postoperative days including PRBC, PLT, FFP, fibrinogen concentrate, PCCs, rFVIIa
Perioperative biological hemostasis | Pre-inclusion - Day 5
  Coagulation tests (PT, aPTT, fibrinogen level) preoperatively, at the end of the surgery (+ thrombin time or ACT ), at arrival in ICU and at POD1, 3 and 5
Complete blood count | Pre-inclusion - Day 5
  Complete blood count preoperatively, at the end of the surgery, at arrival in ICU and at POD1, 3 and 5.
ICU and hospital length of stay | End of study or early termination- Day 30
  calculated ICU and hospital free days
Early postoperative morbidity within 30 postoperative days | Day 30
  Cardiovascular: need for inotropes and/or vasopressors intravenous infusion >24 hours, need for short-term mechanical circulatory support, occurrence of atrial fibrillation and/or ventricular fibrillation/tachycardia, high grade atrioventricular bloc, myocardial infarction, tamponade, symptomatic thromboembolic events.
  Respiratory: duration of mechanical ventilation, re-intubation, ARDS according the Berlin criteria, need for VV ECMO Renal: Kidney Disease Improving Global Outcomes stage (KDIGO) ≥2; need for renal replacement therapy. Serum electrolytes and renal function preoperatively, at arrival in ICU and at POD1, 3 and 5.
  Neurology: transient and permanent stroke, epilepsy, confusion Infectious: mediastinitis, septic shock, pneumopathy and bacteremia Abdominal: mesenteric ischemia, upper and/or lower gastrointestinal bleeding. Liver function tests preoperatively, at arrival in ICU and at POD1, 3 and 5.
  30-day all-cause mortality

OTHER OUTCOMES:
COST-BENEFIT | Day 30 /+2 days
  * Hospital incomes will correspond to the Groupe Homogène de Séjour (GHS) of each patient
  * Hospital expenditure (in-hospital stay, operating room occupancy, transfusions, treatment of infections) valued in the perspective of hospital centers, using data from the national cost studies with common methodology and from analytical accounting.
  * The difference between hospital incomes and hospital expenditures for each patient will be used to estimate the cost-benefit of the filtration-based autotransfusion SAME device as compared to centrifugation-based autotransfusion devices.
Haemoglobin and plasma free haemoglobin | just before surgery as well as 6+/-2 hours after surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: haemoglobin level and plasma free haemoglobin will be performed Blood samples will be also collected from the patient just before surgery as well as 6+/-2 hours after surgery to measure plasma free haemoglobin level.
Hematocrit | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: hematocrit level will be performed.
Complete blood count | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: complete blood count will be performed
Unfractionated heparin anti-Xa | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: unfractionated heparin anti-Xa level will be performed
Fibrinogen | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: fibrinogen level will be performed
Triglycerides | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: triglycerides level will be performed
Total proteins | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: total proteins level will be performed
Potassium | During the surgery
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post treatment) during the first two processing cycles.
  - Laboratory analyses: potassium level will be performed
Blood viscoelasticity assessment | just before and immediately after re-infusion, pré-treatment and just after traitement by the autotransfusion device
  Patients in whom the salvaged blood from mediastinal shed and residual cardiopulmonary bypass circuit volume will be processed and not reinfused before protamine infusion will be included in this ancillary study.
  Blood samples will be collected from the patient just before and immediately after re-infusion of the processed blood and sent to the haematology laboratory to perform viscoelasticity assessment Quantra QPlus™
Complete bloof count | just before and immediately after re-infusion, pré-treatment and just after traitement by the autotransfusion device
  Patients in whom the salvaged blood from mediastinal shed and residual cardiopulmonary bypass circuit volume will be processed and not reinfused before protamine infusion will be included in this ancillary study.
  Blood samples will be collected from the patient just before and immediately after re-infusion of the processed blood and sent to the haematology laboratory to complete blood count.
INF-γ profiling by mass cytometry CyTOF | just before surgery, one day after surgery, pré-treatment and just after treatment by the autotransfusion device
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post-treatment) during the first cycle of processing for immunology assessment (immune profiling by mass cytometry CyTOF).
  Blood samples will be also collected from the patient for INF-γ assessment (by mass cytometry CyTOF) immediately just before surgery as well as one day after surgery
IL-1β-γ profiling by mass cytometry CyTOF | just before surgery, one day after surgery, pré-treatment and just after treatment by the autotransfusion device
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post-treatment) during the first cycle of processing for immunology assessment (immune profiling by mass cytometry CyTOF).
  Blood samples will be also collected from the patient for IL-1β assessment (by mass cytometry CyTOF) immediately just before surgery as well as one day after surgery
Il-6 profiling by mass cytometry CyTOF | just before surgery, one day after surgery, pré-treatment and just after treatment by the autotransfusion device
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post-treatment) during the first cycle of processing for immunology assessment (immune profiling by mass cytometry CyTOF).
  Blood samples will be also collected from the patient for Il-6 assessment (by mass cytometry CyTOF) immediately just before surgery as well as one day after surgery
IL-8 profiling by mass cytometry CyTOF | just before surgery, one day after surgery, pré-treatment and just after treatment by the autotransfusion device
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post-treatment) during the first cycle of processing for immunology assessment (immune profiling by mass cytometry CyTOF).
  Blood samples will be also collected from the patient for IL-8 assessment (by mass cytometry CyTOF) immediately just before surgery as well as one day after surgery
IL-10 profiling by mass cytometry CyTOF | just before surgery, one day after surgery, pré-treatment and just after treatment by the autotransfusion device
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post-treatment) during the first cycle of processing for immunology assessment (immune profiling by mass cytometry CyTOF).
  Blood samples will be also collected from the patient for IL-10 assessment (by mass cytometry CyTOF) immediately just before surgery as well as one day after surgery
TNFα profiling by mass cytometry CyTOF | just before surgery, one day after surgery, pré-treatment and just after treatment by the autotransfusion device
  Blood samples will be collected from the collection reservoir (pre-treatment) of the autotransfusion device and from the reinfusion bag (post-treatment) during the first cycle of processing for immunology assessment (immune profiling by mass cytometry CyTOF).
  Blood samples will be also collected from the patient for TNFα assessment (by mass cytometry CyTOF) immediately just before surgery as well as one day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Ouattara, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (10):
- France (10):
  - CHU de Bordeaux, Hôpital cardiologique Haut Lévêque - GH Sud, Service Anesthésie Réanimation Cardiovasculaire, Bordeaux, France
  - HOSPICES CIVILS DE LYON, Hôpital Louis Pradel, Service Anesthésie Réanimation, Bron
  - CHU MONTPELLIER, Hôpital Arnaud de Villeneuve, Service Anesthésie Réanimation Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Service Anesthésie Réanimation de chirurgie cardiaque, Nantes
  - Groupe Hospitalier Pitié Salpêtrière, APHP, Service Anesthésie Réanimation chirurgicale, Paris
  - Hôpital Bichat-Claude Bernard, APHP, Service Anesthésie Réanimation, Paris
  - Hôpital Européen Georges Pompidou, AP-HP, Service Anesthésie Réanimation, Paris
  - CHU Rennes, Hôpital Pontchaillou, Service Anesthésie Réanimation 3-Réanimation CTCV, Rennes
  - CHRU STRASBOURG, Nouvel Hôpital Civil, Service Anesthésie Réanimation chirurgicale, Strasbourg
  - CHU Toulouse, Hôpital Rangueil, Service Anesthésie, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon reasonable request to qualified researchers, following review and approval by the study sponsor and ethics committee.

REFERENCES:
- [Derived] Beurton A, Mansour A, Benard A, Pernot M, Brett VE, Batsale C, Aitgougam A, Cordon A, Mouton C, Fresselinat A, Robert G, Imbault J, Nesseler N, Ouattara A. Centrifugation versus filtration-based cell salvage: impact on perioperative bleeding in cardiac surgery-the COLTRANE randomised clinical trial - study protocol. BMJ Open. 2025 Jul 16;15(7):e099423. doi: 10.1136/bmjopen-2025-099423. PMID 40669902